CLINICAL TRIAL: NCT05210608
Title: Remember to Abstain: Assessment of Working Memory Training on Delay Discounting in Low-SES Cigarette Smokers
Brief Title: Working Memory Training on Delay Discounting Among Cigarette Smokers
Acronym: RTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00147684; 5KL2TR002367-05 (NIH)
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Use Disorder/Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Working Memory Training + Behavioral Intervention (Experimental): Participants will complete 10 sessions of a Working Memory Training. All participants will receive behavioral activation (a behavioral intervention for smoking cessation) and nicotine patches.
  Interventions: Behavioral: Working Memory Training + Behavioral Intervention

INTERVENTIONS:
Behavioral: Working Memory Training + Behavioral Intervention — Participants will be randomized to complete 10 sessions of a Working Memory Training. All participants will receive behavioral activation (a behavioral intervention for smoking cessation) and nicotine patches.

SUMMARY:
Despite widespread awareness of significant negative health consequences, cigarette smoking remains the leading cause of preventable morbidity and mortality in the US (Creamer et al., 2019; Jamal, 2018). Moreover, the highest rate of smoking and heaviest burden of smoking-related illness occurs among low-socioeconomic status (SES) individuals relative to higher SES groups (Businelle et al., 2010; Clegg et al., 2009). Low SES individuals are also 40% less likely to succeed in quitting smoking when they attempt to do so (National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health, 2014). One potential explanation for the disparity in rate of smoking and successful quit attempts may be differences in individual rates of delay discounting (DD), i.e., the degree to which rewards loses their value as the delays to their receipt increase (Odum, 2011). A proposed way to reduce steep DD and, potentially, substance use has been computer training for working memory, which has shown favorable results in a sample of individuals with stimulant dependence (Bickel et al., 2011) and substance use broadly (Felton et al., 2019), with the latter even showing decreases in cigarette smoking in a subset of the sample.

DETAILED DESCRIPTION:
The highest rate of smoking and heaviest burden of smoking-related illness occurs among low-SES individuals (Businelle et al., 2010; Clegg et al., 2009). One explanation for this disparity may be differences in individual rates of DD, which have been showed to be reduced with working memory training. (Bickel et al., 2011; Felton et al., 2019). Given the low cost of administering working memory training, such an intervention may be favorable for low-SES populations to improve smoking cessation outcomes.

DD has significant associations with:

Cigarette smoking (smokers tend to have higher rates of DD compared to non-smokers; Bickel et al., 1999);

Smoking treatment outcome (individuals who remained smoke free after a smoking cessation intervention had lower DD compared to those who didn't; González-Roz et al., 2019; Krishnan-Sarin et al., 2007; MacKillop & Kahler, 2009; Yoon et al., 2007); SES (individuals with lower education and income have higher DD rates compared to those who are more educated and affluent; de Wit et al., 2007; Reimers et al., 2009).

An innovative way to reduce DD that has been proposed is via working memory (WM) training. WM refers to one's capacity to hold information while engaging in complex mental tasks, including reasoning, comprehension, and learning (Baddeley, 2010). Previous research has shown that DD and WM correlate negatively (Shamosh et al., 2008), that individuals with higher DD rates show neural deficits in WM (Herting et al., 2010), and that acute nicotine abstinence is associated with WM deficits (Mendrek et al., 2006; Patterson et al., 2010). Furthermore, previous studies targeting WM to reduce DD have shown favorable results in a sample of individuals with stimulant dependence (Bickel et al., 2011) and substance use broadly (Felton et al., 2019), with the latter even showing decreases in cigarette smoking in a subset of the sample.

Although previous research has shown WM training to reduce DD (which would support H3), and cigarette use in a small subsample, the hypotheses of this study are largely exploratory. However, given the theoretical connections between DD, SES, and WM, it is expected that the hypotheses of this project will be supported.

The performance of this project may advance our knowledge of the relevant clinical targets for smoking cessation in low-SES individuals. In particular, this project is expected to shed light on DD as the putative mechanism in smoking for low-SES individuals and the durability of reductions in smoking as a result of reductions in DD through WM training.

Despite the evidence for some successful techniques for reducing DD, little of this work has been translated into intervention approaches to target clinical outcomes. This application seeks to capitalize on the emerging literatures indicating (1) WM training may be an effective and efficient way to reduce DD, and (2) DD is associated with SES, cigarette smoking, and treatment outcomes. Though WM training has been successfully implemented in laboratory-controlled experiments to reduce DD, we are not aware of any interventions for clinical disorders that specifically seek to do so and potentially enhance treatment outcomes.

The development of effective, theoretically coherent interventions addressing cigarette smoking is imperative, particularly interventions that would be feasible, efficacious, and acceptable in low-SES individuals. The proposed research is an innovative approach that capitalizes on previous findings showing reductions in delay discounting and even cigarette smoking. If working memory training is found to improve smoking cessation outcomes as a function of reductions in delay discounting, the project results could be helpful in future development of low-cost interventions for cigarette smoking.

ELIGIBILITY:
Inclusion criteria: To be included in this study, a participant must be 18 years of age or older, who have smoked at least four cigarettes per day for at least 6 months, are interested in quitting cigarette smoking, are at or below the federal poverty line based on persons in family/household and annual household income:

* 1 -- $12,880
* 2 -- $17,420
* 3 -- $21,960
* 4 - $26,500
* 5 -- $31,040
* 6 -- $35,580
* 7 -- $40,120
* 8 -- $44,660
* 9 - add $4,540 for each additional person,

OR they or their child(ren) utilize a federal program for low-income individuals, and are willing to participate in a 5-week working memory training program as a pretreatment adjunct to behavioral group + nicotine replacement therapy (NRT; via nicotine patches).

Exclusion criteria: Participants must not indicate a severe substance use disorder according to the DSM-V with any substance other than tobacco or have any significant medical or psychiatric condition. Such conditions could include traumatic brain injury, dementia, significant learning disability, or psychotic symptoms. Participants must be at least at a 5th-grade reading level. In case that participants are excluded, they will be provided with resources in the community and provided with contact information for the Kansas Tobacco Quitline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Collado, Principal Investigator — KU-Lawrence
Locations (1):
- Swope Health Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Working Memory Training + Behavioral Intervention
Started | 13
Completed | 8
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Working Memory Training+ Behavioral Intervention: Participants will complete 10 sessions of a Working Memory Training. All participants will receive behavioral activation (a behavioral intervention for smoking cessation) and nicotine patches.
Arm/Group | Working Memory Training+ Behavioral Intervention
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.37 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Delay Discounting (DD) Measure [Mean (Full Range); unit: k-value] — DD was assessed using a computerized binary choice task where participants chose between an immediate sum and a larger delayed sum (1 day to 25 years). A computerized algorithm adjusted the immediate reward over 7 trials to determine an indifference point (k) for each amount. DD was calculated for $50, $200, and $1,000. Higher scores indicate greater discounting of delayed rewards. Values near 0 or negative suggest slow discounting, while values above 1 indicate heavy discounting. There is no strict upper or lower limit.
  k-value | -5.21 [-12.12 to -0.19]

OUTCOME MEASURES:

1. Primary Outcome: Delay Discounting
Description: Delay Discounting (DD) was measured via an established computerized binary choice task in which participants choose between an amount of money available immediately and larger amount of money available after a specified delay (1 day to 25 years). A computerized algorithm adjusts the immediately available reward across seven trials to determine an indifference point (k) for each amount/delay pairing. Indifference points are then used to calculate a rate of delay discounting for a $50, $200, $1,000 "larger later" sum. Larger scores mean greater delay discounting. While there is no strict minimum or maximum k-value, but in practical research settings, typical k-values often range from close to 0 for individuals who discount delayed rewards very slowly to values above 1 for those who heavily discount delayed rewards. There is no strict lower or upper bound, but values can be extremely high (above 1) if an individual very strongly prefers immediate rewards.
Time Frame: Baseline, Post-treatment, 1 month follow up
Measure: Mean (95% Confidence Interval); unit: k-value
Arm/Group | Working Memory Training + Behavioral Intervention
Number analyzed (Participants) | 13
k-value
  Baseline | -5.21 [-12.12 to -0.19]
  Post-treatment | -6.57 [-10.66 to -4.24]
  1 month follow up | -7.13 [-10.19 to -4.15]
Statistical Analysis 1: Comparison: Working Memory Training + Behavioral Intervention; We analyzed whether significant changes occurred between baseline and the post-treatment assessment; Test type: Superiority; p = .29, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [-.85 to 2.18], Standard Error of Mean .55
Statistical Analysis 2: Comparison: Working Memory Training + Behavioral Intervention; We analyzed whether significant changes occurred between baseline and the 1 month follow up; Test type: Superiority; p = .48, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 1.92, 95% CI 2-sided [-3.45 to 5.79], Standard Error of Mean 1.45

2. Primary Outcome: Timeline Follow-Back (TLFB): Number of Total Cigarettes Smoked Per Week
Description: The Timeline Follow-Back (TLFB) for cigarette smoking is a self-report method used to assess an individual's smoking behavior over a specified period and specified as one week for this study. In this method, individuals are guided to recall their daily cigarette use by referencing events, routines, and cues that help them accurately track their smoking patterns. They are asked to document the number of cigarettes smoked each day, which provides a detailed, day-by-day account of their smoking habits. This data was then be summed to give a weekly total cigarettes smoked per week. The TLFB approach is valued for its reliability and ability to capture fluctuations in smoking behavior over time.
Time Frame: Baseline, Post-treatment, 1 month follow up
Measure: Mean (Standard Deviation); unit: number of total cigarettes/week
Arm/Group | Working Memory Training+ Behavioral Intervention
Number analyzed (Participants) | 13
number of total cigarettes/week
  Baseline | 76.53 (60.70)
  Post-treatment | 38.83 (40.15)
  1 month follow up | 59.50 (27.55)
Statistical Analysis 1: Comparison: Working Memory Training+ Behavioral Intervention; We analyzed whether there were significant differences in number of total cigarettes smoked per week from baseline to Post-treatment; Test type: Superiority; p = 0.015, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 37.7, 95% CI 2-sided [19.90 to 102.10], Standard Error of Mean 14.80
Statistical Analysis 2: Comparison: Working Memory Training+ Behavioral Intervention; We analyzed whether there were significant differences in number of total cigarettes smoked per week from baseline to 1 month follow-up; Test type: Superiority; p = .08, t-test, 2 sided; Mean Difference (Final Values) = 17.03, 95% CI 2-sided [-14.57 to 142.57], Standard Error of Mean 24.69

3. Primary Outcome: Carbon Monoxide Levels
Description: Participant reports of abstinence will be verified by expired carbon monoxide (< 6 ppm cutoff for stated abstinence). CO levels are collected via a CO monitor.
Time Frame: Baseline, Post-treatment, 1 month follow up
Measure: Mean (Standard Deviation); unit: ppm (parts per million)
Arm/Group | Working Memory Training+ Behavioral Intervention
Number analyzed (Participants) | 13
ppm (parts per million)
  Baseline | 17.70 (11.65)
  Post-treatment | 17.67 (9.44)
  1 month follow up | 30 (17.45)
Statistical Analysis 1: Comparison: Working Memory Training+ Behavioral Intervention; We analyzed whether there were significant differences in carbon monoxide ppm from baseline to Post-treatment; Test type: Superiority; p = .90, t-test, 2 sided; Mean Difference (Final Values) = .03, 95% CI 2-sided [-9.86 to 8.86], Standard Error of Mean 3.64
Statistical Analysis 2: Comparison: Working Memory Training+ Behavioral Intervention; We analyzed whether there were significant difference in carbon monoxide ppm from baseline to the 1 month follow-up; Test type: Superiority; p = .32, t-test, 2 sided; Mean Difference (Final Values) = -12.30, 95% CI 2-sided [-49.42 to 22.42], Standard Error of Mean 11.29

4. Primary Outcome: Working Memory
Description: Working memory was assessed by adding the scores of 3 different working memory measures: 1) the total achievement score in the Tower of Hanoi, 2) the total recall score of the Hopkins Verbal Learning Test- Revised and 3) the total scaled score of the Letter Number Sequencing. These measures are commonly used to assess working memory. In this study, the composite score of all measures ranged between 36 and 89 with higher scores representing greater working memory,
Time Frame: Baseline, Post-treatment, 1 month follow up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Working Memory Training+ Behavioral Intervention
Number analyzed (Participants) | 13
Scores on a scale
  Baseline | 58.61 (14.43)
  Post-treatment | 61.33 (11.13)
  1 month follow up | 71.25 (13.42)
Statistical Analysis 1: Comparison: Working Memory Training+ Behavioral Intervention; We analyzed whether there were significant differences in working memory scores from baseline to post-treatment; Test type: Superiority; p = .18, t-test, 2 sided; Mean Difference (Final Values) = -2.72, 95% CI 2-sided [-5.10 to 19.10], Standard Error of Mean 4.36
Statistical Analysis 2: Comparison: Working Memory Training+ Behavioral Intervention; We analyzed whether there were significant differences in working memory scores from baseline to the 1 month follow up; Test type: Superiority; p = .18, t-test, 2 sided; Mean Difference (Final Values) = -12.64, 95% CI 2-sided [-25.38 to 7.38], Standard Error of Mean 5.14

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events, or Other Adverse Events, were not monitored or assessed
Description: All-Cause Mortality, Serious Adverse Events, or Other Adverse Events, were not monitored or assessed
Arm/Group | Working Memory Training + Behavioral Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT05210608/Prot_SAP_000.pdf